CLINICAL TRIAL: NCT01368965
Title: Evaluation of the Ulthera® System for Obtaining Lift and Tightening of the Cheek Tissue and Improvement in Jawline Definition and Submental Skin Laxity in Patients With Fitzpatrick Skin Phototypes 3 Through 6
Brief Title: Lifting and Tightening of the Face in Subjects With Skin of Darker Color
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ULT-112
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Facial Skin Laxity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ulthera® System treatment (Experimental)
  Interventions: Device: Ulthera® System treatment

INTERVENTIONS:
Device: Ulthera® System treatment — Ulthera® System treatment delivering focused ultrasound energy

SUMMARY:
This prospective, multi-center, single treatment clinical trial evaluates the clinical outcomes associated with non-invasive treatment to obtain lift and tightening of facial tissue and improve jawline definition in subjects with darker skin color utilizing the Ulthera® System to deliver focused ultrasound energy below the skin surface.

DETAILED DESCRIPTION:
The primary objective of this clinical trial is to demonstrate the effectiveness of the Ulthera® System for the non-invasive treatment to obtain overall lift and tightening of facial tissue and jawline definition improvement.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 30 to 65 years.
* Subject in good health.
* Subjects who desire lift and tightening of cheek tissue, improvement in jawline definition and/or submental skin laxity.
* Fitzpatrick skin phototypes of 3 through 6.
* Provide written informed consent and HIPAA authorization

Exclusion Criteria:

* Pregnant or lactating.
* Presence of an active systemic or local skin disease that may affect wound healing.
* Severe solar elastosis.
* Excessive subcutaneous fat on the cheek.
* Excessive skin laxity on the lower face and neck.
* Significant scarring in areas to be treated.
* Significant open facial wounds or lesions.
* Severe or cystic acne on the face.
* Presence of a metal stent or implant in the facial area to be treated.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-03; Primary Completion 2011-10 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hema Sundaram, M.D., Principal Investigator — Dermatology, Cosmetic & Laser Surgery; Monte O Harris, M.D., Principal Investigator — Harris Aesthetics, LLC
Locations (2):
- United States (2):
  - Harris Aesthetics, LLC, Chevy Chase, Maryland
  - Dermatology, Cosmetic & Laser Surgery, Rockville, Maryland

REFERENCES:
- [Derived] Harris MO, Sundaram HA. Safety of Microfocused Ultrasound With Visualization in Patients With Fitzpatrick Skin Phototypes III to VI. JAMA Facial Plast Surg. 2015 Sep-Oct;17(5):355-7. doi: 10.1001/jamafacial.2015.0990. PMID 26313402

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects desiring lift/tightening of cheek tissue, or improved jawline definition and/or submental skin laxity, and were Fitzpatrick skin types 3-6 were recruited. Fifty-four subjects were enrolled at two facilities. Study recruitment initiated 2/16/11; follow-up concluded 1/18/12.
Pre-assignment Details: Fifty-four subjects who met study eligibility requirements were assigned a study subject ID. Two subjects withdrew from the study due prior to study treatment. Data from these subjects are not included in the demographic summaries or in the efficacy analyses. Fifty-two subjects received study treatment.
Groups:
- Treated Subjects: All treated study subjects received a full face Ulthera® treatment.
Period: Overall Study
Arm/Group | Treated Subjects
Started | 52 (Two subjects withdrew consent prior to study treatment. Data analyses are based on 52 subjects.)
Subject Withdrawal Prior to Treatment | 2
Completed | 40
Not Completed | 12
Not completed — Lost to Follow-up | 12

BASELINE CHARACTERISTICS:
Population: Fifty-four subjects were consented and enrolled. Two subjects withdrew consent prior to treatment. Data analyses are based on 52 treated subjects.
Groups:
- Treated Subjects: Study subjects who received a full face Ulthera treatment. (n=52)
Arm/Group | Treated Subjects
Number analyzed (Participants) | 52
Age, Continuous [Mean (Full Range); unit: years] | 53 [32 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 1
Race/Ethnicity, Customized [Number; unit: participants]
  African American/Black | 35
  Hispanic/Latino | 5
  Asian | 10
  Other | 2
Region of Enrollment [Number; unit: participants]
  United States | 52
Fitzpatrick Skin Type [Number; unit: participants] — Skin Type I = White;very fair,red or blonde hair blue eyes;freckles;Always burns, never tans
  Skin Type II = White, fair, red or blond hair; blue, hazel or green eyes;Usually burns, tans with difficulty
  Skin Type III = Cream white; fair with any eye or hair color (common); Sometimes mild burn, gradually tans
  Skin Type IV = Brown; typical Mediterranean Caucasian skin; Rarely burns, tans with ease
  Skin Type V = Dark Brown; mid-eastern skin types; Very rarely burns, tans easily
  Skin Type VI = Black; Never burns, tans very easily
  participants
    Type III | 9
    Type IV | 25
    Type V | 15
    Type VI | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Overall Lifting and Tightening of Treated Tissue
Description: The percentage of participants assessed to have improvement in skin laxity, i.e., lifted and tightened skin in the areas treated with the Ulthera System, as determined by three masked assessors comparing pre-treatment and 90-days post-treatment photos
Time Frame: 90 days post treatment
Population: Masked, qualitative assessment of standardized photographs at 90 days post treatment compared to baseline, could not be completed as images taken at one site were not recovered due to poor data management and staffing issues at the site.
Arm/Group | Treated Subjects
Number analyzed (Participants) | 0

2. Secondary Outcome: Global Aesthetic Improvement at 90 Days Post-treatment
Description: At 90 days post-treatment, each site investigator and each subject completed a Global Aesthetic Improvement Scale (GAIS), comparing with pre-treatment photos. PGAIS = Physician Global Aesthetic Improvement Scale; SGAIS = Subject Global Aesthetic Improvement Scale.
Time Frame: 90 Days post-treatment
Population: The GAIS is 5-point scale (1-5) describing an overall assessment as follows:
  1. = Very Much Improved
  2. = Much Improved
  3. = Improved
  4. = No Change
  5. = Worse
Measure: Number; unit: percentage of participants improved
Arm/Group | Treated Subjects
Number analyzed (Participants) | 48
percentage of participants improved
  PGAIS - Improved to Very Much Improved | 85.4
  SGAIS - Improved to Very Much Improved | 79.2

3. Secondary Outcome: Global Aesthetic Improvement at 180 Days Post-treatment
Description: At 180 days post-treatment, each site investigator and each subject completed a Global Aesthetic Improvement Scale (GAIS), comparing with pre-treatment photos. PGAIS = Physician Global Aesthetic Improvement Scale; SGAIS = Subject Global Aesthetic Improvement Scale.
Time Frame: 180 days post-treatment
Population: Subjects completing the 180-Day SGAIS = 39; however, the 180-Day PGAIS was not obtained for 2 subjects. PGAIS data are based on n=37.
  The GAIS is 5-point scale (1-5) describing an overall assessment as follows:
  1. = Very Much Improved
  2. = Much Improved
  3. = Improved
  4. = No Change
  5. = Worse
Measure: Number; unit: percentage of participants improved
Arm/Group | Treated Subjects
Number analyzed (Participants) | 39
percentage of participants improved
  PGAIS - Improved to Very Much Improved | 54.0
  SGAIS - Improved to Very Much Improved | 77.0

4. Secondary Outcome: Patient Satisfaction Questionnaire
Description: Subjects indicated whether they saw improvement, i.e., providing a Yes/No response, in face and neck characteristics at three months (D90) post Ulthera treatment. Pre-treatment and Day 90 post-treatment photographs were available for viewing during the assessment. Subjects also had a mirror in hand for real time assessment. Subjects' Yes/No responses were tabulated.
Time Frame: 90 Days post-treatment
Population: Data analyzed includes PSQ responses at 90 days post-treatment assessing subjects' satisfaction with study treatment. Responses were tabulated. Outcomes reported represent the percentage of subjects reporting any satisfaction, i.e., Very Satisfied and Satisfied.
Measure: Number; unit: percentage of participants Satisfied
Arm/Group | Treated Subjects
Number analyzed (Participants) | 47
percentage of participants Satisfied | 83.0

5. Secondary Outcome: Patient Satisfaction Questionnaire
Description: Subjects indicated whether they saw improvement, i.e., providing a Yes/No response, in face and neck characteristics at six months (D180) post Ulthera treatment. Pre-treatment and Day 180 post-treatment photographs were available for viewing during the assessment. Subjects also had a mirror in hand for real time assessment. Subjects' Yes/No responses were tabulated.
Time Frame: 180 days post-treatment
Population: Data analyzed includes PSQ responses at 180 days post-treatment assessing subjects' satisfaction with study treatment. Responses were tabulated. Outcomes reported represent the percentage of subjects reporting any satisfaction, i.e., Very Satisfied and Satisfied.
Measure: Number; unit: percentage of participants Satisfied
Arm/Group | Treated Subjects
Number analyzed (Participants) | 40
percentage of participants Satisfied | 72.5

6. Other Pre Specified Outcome: Subject Assessment of Pain
Description: Subject assessment of pain using a validated Numeric Rating Scale (NRS), 0-10, where 0 = no pain and 10=worse pain possible. Subjects' sensory responses to the treatment exposures were recorded using the NRS for each anatomical region.
Time Frame: During Ulthera treatment
Measure: Mean (Full Range); unit: Average NRS score
Arm/Group | Treated Subjects
Number analyzed (Participants) | 52
Average NRS score
  Submental Region | 6 [2 to 10]
  Submandibular Region | 6 [2 to 10]
  Cheek Region | 6 [1 to 10]

ADVERSE EVENTS:
Groups:
- Enrolled Subjects: Includes all subjects enrolled, including 52 treated subjects and 2 non-treated subjects who withdrew consent prior to treatment.
Arm/Group | Enrolled Subjects
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 0/54

LIMITATIONS AND CAVEATS:
Study Limitations:

* Masked assessment was not completed as photos were not usable, i.e., poor image quality, positioning and timing.
* Site staffing changes.
* Overburdened site staff.
* Poor photography quality
* Subject selection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No